CLINICAL TRIAL: NCT03725592
Title: Participatory Interventions to Reduce Arsenic Exposure in American Indian Communities
Brief Title: Strong Heart Water Study
Acronym: SHWS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Columbia University (Other); Missouri Breaks Industries Research, Inc. (Other); National Institute Of Allergy & Infectuous Disease (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00006504
Record Dates: First submitted 2018-07-06; First posted 2018-10-31 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Arsenic Poisoning
Keywords: arsenic; drinking water
MeSH Terms: conditions — Arsenic Poisoning

STUDY DESIGN:
Intervention Model Description: Recruit and prospectively follow 300 households and 600 participants (2 per household) to one of 2 study arms (150 households per arm). Each arm will receive arsenic removal devices. However the Standard Arm will only be provided with written instructions on how to use the arsenic removal device and follow-up phone calls, while the Intensive Education Arm will receive up to 5 additional in-visits and phone calls to provide support regarding the health implications of arsenic and the proper use and maintenance of the arsenic removal device.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Treatment (Active Comparator): Receives arsenic removal device and written instructions and phone calls on how to use the device (Arsenic Removal Device)
  Interventions: Other: Standard Treatment
- Intensive Education (Experimental): Receives the Standard Treatment plus in-person visits and phone calls for follow-up (Community Participatory Arsenic Mitigation)
  Interventions: Other: Standard Treatment; Behavioral: Intensive Education

INTERVENTIONS:
Other: Standard Treatment — Participant households receive a point of use arsenic removal device and a replacement filter. Households are also provided with an instruction manual on how to use the device.
  Other Names: Arsenic Removal Device
Behavioral: Intensive Education — Participant households receive up to five additional in-person visits and phone calls to provide support regarding the health implications of arsenic and the proper use and maintenance of the arsenic removal device.
  Other Names: Community Participatory Arsenic Mitigation
  Arms: Intensive Education

SUMMARY:
Develop and evaluate the effectiveness of multi-level participatory interventions in reducing arsenic exposure among American Indian (AI) communities from North and South Dakota who participated in the Strong Heart Study (SHS).

DETAILED DESCRIPTION:
Design, implement, and evaluate multi-level participatory interventions that can lead to a sustained reduction in arsenic exposure in adults and children in Cheyenne River, Oglala, and Spirit Lake communities in North/South Dakota by: 1) building local capacity at the tribal and community levels to ensure the long-term sustainability of the interventions. 2) conduct a 2-arm cluster-randomized controlled trial comparing arsenic removal device only to removal device and intensive education and promotion among 300 households, 600 participants.

ELIGIBILITY:
Inclusion Criteria:

* Arsenic levels in household drinking water must be ≥10 µg/L
* Households must have ≥1 adult ≥18 years of age eligible and willing to participate.
* Household must have an active well on the property that is used for drinking water.
* Household must have indoor plumbing and a permanent heat source.
* Participant must plan to reside in the household for the next year, must reside in the residence for ≥4 days/week, and year round (i.e. all seasons).
* ≥1 household members must identify as American Indian.
* Household must be willing to grant study members access to the interior of their household for screening and data collection.

Exclusion Criteria:

* Arsenic levels in household drinking water <10 µg/L
* Households with no adult ≥18 years of age eligible and willing to participate.
* Households without an active well on the property that is used for drinking water (i.e. connected to municipal water supply).
* Households without indoor plumbing and/or a permanent heat source.
* Participant planning to reside in the household <1 year, residing in the residence for <4 days/week, or not year round (i.e. not during all seasons).
* No household member identifies as American Indian.
* Household unwilling to grant study members access to the interior of their household for screening and data collection.

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2026-05-04 (Estimated); Study Completion 2026-05-04 (Estimated)

PRIMARY OUTCOMES:
Urine arsenic concentrations in household members | 6 months post-installation of the arsenic removal device
  (1a) urine arsenic concentrations among household members (in parts per billion, µg/L)

SECONDARY OUTCOMES:
Arsenic concentrations in filtered water | 6 months post-installation of the arsenic removal device
  (2a) water arsenic concentrations from arsenic removal device (parts per billion, µg/L)
Water usage from arsenic removal device | 6 months post-installation of the arsenic removal device
  (2b) water usage from removal device (from flow meter, in gallons)
Biomarkers of cardiovascular disease | 6 months post-installation of the arsenic removal device
  (2c) biomarkers of cardiovascular disease (soluble adhesion molecules) in household members
Biomarkers of diabetes | 6 months post-installation of the arsenic removal device
  (2d) biomarkers of diabetes (hemoglobin A1c) in household members
Biomarkers of pulmonary function | 6 months post-installation of the arsenic removal device
  (2e.1) lower forced expiratory volume in 1 second (FEV1) (actual performance in liters of air, percent of predicted values)
Biomarkers of pulmonary function | 6 months post-installation of the arsenic removal device
  (2e.2) lower forced vital capacity (FVC) among household members (actual performance in liters of air, percent of predicted values)
Blood pressure | 6 months post-installation of the arsenic removal device
  (2f) systolic and diastolic blood pressure levels
Long-term urine arsenic concentrations in household members | 1 year post-installation of the arsenic removal device
  (2g) long-term sustainability assessment to evaluate arsenic concentrations in urine among household members (parts per billion, µg/L)
Long-term functionality of arsenic removal device | 1 year post-installation of the arsenic removal device
  (2h) long-term sustainability assessment to evaluate water arsenic concentrations from arsenic removal device (parts per billion, µg/L)
Long-term water usage from arsenic removal device | 1 year post-installation of the arsenic removal device
  (2i) long-term sustainability assessment to evaluate water usage from removal device (from flow meter, in gallons)
Long-term maintenance of arsenic removal device | 1 year post-installation of the arsenic removal device
  (2j) long-term sustainability assessment to evaluate self-reported maintenance of the arsenic removal device (Did household change the device filter when indicated by light on spigot? Does household have replacement filter(s) available for subsequent filter change(s)?)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Marie George, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, ICTR, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Endres K, Zacher T, Richards F, Bear Robe L, Powers M, Yracheta J, Harvey D, Best LG, Red Cloud R, Black Bear A, Ristau S, Aurand D, Skinner L, Perin J, Cuny C, Gross M, Thomas ED, Rule A, Schwab K, Moulton LH, O'Leary M, Navas-Acien A, George CM. Behavioral determinants of arsenic-safe water use among Great Plains Indian Nation private well users: results from the Community-Led Strong Heart Water Study Arsenic Mitigation Program. Environ Health. 2023 May 15;22(1):42. doi: 10.1186/s12940-023-00965-0. PMID 37183246